CLINICAL TRIAL: NCT01374100
Title: Effect of Qigong Therapy in Patients With Advanced NSCLC and GI Cancer Undergoing Chemotherapy
Brief Title: Effect of Qigong Therapy in Patients With Advanced Lung and Gastrointestinal Cancer Undergoing Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual, and revised power calculation for primary end-points
Sponsor: McGill University (Other)
Collaborators: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Thomas Jagoe, Associate Professor of Medicine, McGill University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 08-068
Record Dates: First submitted 2011-04-13; First posted 2011-06-15 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Cancer of the Gastrointestinal Tract
Keywords: Qigong; Complementary Medicine; Exercise; Traditional Chinese Medicine; Meditation; Standard Exercise; Chemotherapy; Advanced cancer; Quality of Life; Functional Assessment of Cancer Therapy; Hospital Anxiety and Depression Scale; Anxiety; Depression; Cancer Nutrition-Rehabilitation Program; Edmonton Symptom Assessment Scale; Simmonds Functional Assessment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Gastrointestinal Neoplasms; Motor Activity; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Exercise (Active Comparator): See methods below - standard strength and endurance training
  Interventions: Behavioral: Standard Exercise; Behavioral: Qigong Exercise
- Qigong exercise (Experimental): See methods below - medical QiGong therapy session
  Interventions: Behavioral: Standard Exercise; Behavioral: Qigong Exercise

INTERVENTIONS:
Behavioral: Standard Exercise — The standard exercise therapy program will include 12 treatments of approximately 45 minutes duration, twice a week for a period of six weeks by the same instructor and at the same location as for Qigong therapy. This exercise program is supervised and consists of cardio-vascular and resistance training exercises. Participants are asked to refrain from practicing Qigong during this 6 week period.
Behavioral: Qigong Exercise — Qigong therapy will be led by a trained Qigong instructor and will occur for 45 minutes sessions, twice a week for a period of six weeks. Qigong is a self-directed walking exercise program that involves arm movements that are coordinated with slight movements of the waist, while in a state of deep relaxation or meditation. Patients will be asked to refrain from independent resistance or cardiovascular training during this 6 week period.

SUMMARY:
Cancer patients face a number of symptoms related to treatment or disease which may impair quality of life, such as decreased functional capacity, fatigue, nausea an vomiting, distress, depression and unmet psychological needs. Due to this array of symptoms, cancer patients often seek supportive complementary and alternative medicine, which many patients use along with conventional treatments. Qigong, a type traditional chinese medicine, is a mind-body exercise that combines meditation, slow physical movements, and controlled breathing. The investigators hypothesise that Qigong therapy is better in the reduction of anxiety and depression levels and the improvement of quality of life in patients with lung and gastrointestinal (GI) cancer who are eligible for anti-cancer treatment, when compared to standard exercise training.

DETAILED DESCRIPTION:
As per summary above

ELIGIBILITY:
Inclusion Criteria:

1. A pathologically (histological or cytological) confirmed clinical diagnosis of non-small cell lung cancer (NSCLC) or GI cancer
2. Stage 3 or 4 disease and eligible for anti-cancer treatment
3. Performance status (PS) of 0 - 2 as determined by the Eastern Cooperative Oncology Group-Performance Status
4. Life expectancy estimated at > 4 months
5. Age 18 years or older
6. Willing and able to provide informed consent
7. Must be approved for participation by the oncology treatment team
8. Able to communicate in French or English

Exclusion Criteria:

1. Contraindication to exercise as determined by the oncology treatment team
2. Severe cardiac or neuro-muscular/skeletal disease
3. Engaging in interventions to address anxiety or depressive symptoms
4. Brain metastases
5. Active psychiatric conditions
6. Pregnant or breast-feeding mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in Depression and Anxiety | 6 weeks
  Depression and anxiety will be measured using the Hospital Anxiety Depression Scale (HADS); The HADS is a 14-item self-rated questionnaire, consisting of two 7-item subscales. It was developed to identify anxiety and depression in non-psychiatric medical outpatients. Each item on the HADS is scored from 0 (no problem) to 3 (maximum distress). The HADS will be administered within 2 weeks of completing each exercise program.
Change in Quality of Life (QoL) | 6 weeks
  The general version of the Functional Assessment of Cancer Therapy scale (FACT-G) will be used to measure Quality of Life (QoL) after completion of each 6 week exercise program. This questionnaire consists of 4 subscales: Physical well-being (PWB), Social well-being (SWB), Emotional well-being (EWB) and Functional well-being (FWB). A change of 4 points on the total FACT score is regarded as clinically significant.

SECONDARY OUTCOMES:
Change in functional capacity | 6 weeks
  Functional capcity will be measured using the Simmonds Functional Assessment (SFA) within 2 weeks of finishing each 6-week exercise program. This tool consists of eight items: putting on a sock, tying a belt, putting coins in a cup, reaching forward, repeated reach up (3 times), repeated sit to stand (2 times), speed walk for 50 feet, and walking for 6 minutes. Patient satisfaction will be measured by asking all participants to answer a two item questionnaire with a 10-point visual analog scale response option.
Change in cancer Symptoms | 6 weeks
  Symptoms commonly reported by lung and GI cancer patients will be measured using the Edmonton Symptom Assessment Scale (ESAS). The ESAS is a 12-item patient rated symptom questionnaire scored using a 10-point visual analogue scale. The ESAS will be administered within 2 weeks of completing each 6-week exercise program.
Program Satisfaction | 6 weeks
  Patient satisfaction will be measured by asking all participants to answer a two-item questionnaire after they have completed each 6-week exercise program.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jagoe, MD, PhD, Principal Investigator — McGill, Cancer Nutrition Rehabilitation Program
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Peer-reviewed manuscripts and conference proceedings
Supporting Information: Study Protocol, SAP, CSR
Time Frame: All group data already supplied in published manuscript
Access Criteria: Other specific anonymized data on participants supplied for academic/research purposes by application to the senior author.

REFERENCES:
- [Result] Vanderbyl BL, Mayer MJ, Nash C, Tran AT, Windholz T, Swanson T, Kasymjanova G, Jagoe RT. A comparison of the effects of medical Qigong and standard exercise therapy on symptoms and quality of life in patients with advanced cancer. Support Care Cancer. 2017 Jun;25(6):1749-1758. doi: 10.1007/s00520-017-3579-x. Epub 2017 Jan 19. PMID 28102437